CLINICAL TRIAL: NCT05313737
Title: Opt-in vs. Opt-out Mammography Screening Outreach: a Randomized Controlled Trial
Brief Title: Opt-in vs. Opt-out for Breast Cancer Screening
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: VA Puget Sound Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Alaina Mori, Staff Physician, VA Puget Sound Health Care System
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: MAMMoutreach
Record Dates: First submitted 2022-02-01; First posted 2022-04-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Breast Cancer
Keywords: Cancer Screening; Adherence
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Automated phone opt-in message (Experimental): Audiocare message requiring Veteran to confirm that they would like to participate in screening and have consult sent
  Interventions: Other: Automated message
- Opt-out scheduling (Experimental): Consult automatically sent and Veteran called to schedule screening
  Interventions: Other: Opt-out scheduling

INTERVENTIONS:
Other: Automated message — Automated message via phone call (audiocare)
  Arms: Automated phone opt-in message
Other: Opt-out scheduling — Scheduling via non-automated phone call
  Arms: Opt-out scheduling

SUMMARY:
This is a randomized controlled trial that will evaluate the effectiveness two different outreach strategies for a population-based breast cancer screening program at the VA Puget Sound among average risk female Veterans who are due for breast cancer screening.

DETAILED DESCRIPTION:
This is a prospective, randomized controlled trial that will evaluate the effectiveness of two different outreach strategies in improving adherence to breast cancer screening via mammography.

Average risk female Veterans who are due for breast cancer screening (defined as aged 45-75 with no previous history of bilateral mastectomy, not under hospice care, and alive at the time of screening) will be identified through administrative data.

Veterans eligible for enrollment into the trial will be randomized in a 1:1 allocation using permuted block randomization (with random block sizes of 2 and 4) to the following interventions:

Arm 1: Automated phone opt-in message Intervention Type: Audiocare message requiring Veteran to confirm that they would like to participate in screening and have consult sent Arm 2: Opt-out scheduling Intervention Type: Consult automatically sent and Veteran called to schedule screening

Randomization will be stratified within arms by prior screening status (prior screener vs. never screener).

The study's primary outcome of interest is screening completion at 100 days post randomization. The study's secondary outcome of interest is screening scheduling at 100 days post randomization. Subgroup analysis aim 1 will explore whether the differences in breast cancer screening completion between investigational groups varies according to the Veterans' race/ethnicity. Subgroup analysis aim 2 will explore whether the differences in breast cancer screening scheduling between investigational groups varies according to the Veterans' race/ethnicity. Enrollment in the trial will occur between March 1, 2022 and August 31, 2022.

ELIGIBILITY:
Inclusion Criteria:

* female Veterans aged 45-75
* assigned to a primary care provider at the VA Puget Sound as of January 1, 2022 with at least 1 year of prior data available
* due for breast cancer screening (have not had a mammogram in the last 12 months)

Exclusion Criteria:

* must not be any indication of current receipt of hospice care
* no record of recent death in the administrative data
* not scheduled for either a screening or diagnostic mammogram within the following 12 weeks from assessment.
* not have a personal history of bilateral mastectomy.

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — female only
Enrollment: 871 (Estimated)
Dates: Start 2022-04-18 (Estimated); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of mammograms completed at 100 days post randomization | 100 days post randomization
  Percent of mammograms completed

SECONDARY OUTCOMES:
Percentage of mammograms scheduled at 100 days post randomization | 100 days post randomization
  Percent of mammograms scheduled

OTHER OUTCOMES:
Percentage of mammograms cancelled at 100 days post randomization | 100 days post randomization
  Percent of mammograms cancelled
Percentage of mammograms active at 100 days post randomization | 100 days post randomization
  Percent of mammograms active

CONTACTS AND LOCATIONS:
Overall Officials: Ashok Reddy, MD, Principal Investigator — VA Puget Sound Health Care System; Stefanie Deeds, MD, Principal Investigator — VA Puget Sound Health Care System
Locations (1):
- VA Puget Sound Health Care System, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marcotte LM, Deeds S, Wheat C, Gunnink E, Gray K, Rojas J, Finch C, Nelson K, Reddy A. Automated Opt-Out vs Opt-In Patient Outreach Strategies for Breast Cancer Screening: A Randomized Clinical Trial. JAMA Intern Med. 2023 Nov 1;183(11):1187-1194. doi: 10.1001/jamainternmed.2023.4321. PMID 37695621